CLINICAL TRIAL: NCT00294255
Title: Risperidone Plus Mood Stabilizer in the Treatment of Mixed Mania
Brief Title: Risperidone Plus Mood Stabilizer in Treatment of Mixed Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIS-USA-T290
Record Dates: First submitted 2005-09-13; First posted 2006-02-20 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2013-02

CONDITIONS: Bipolar Disorder
Keywords: mixed mania; depression; irritability
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Risperidone (Experimental): patients will receive risperidone for up to 20 weeks
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — risperidone will be administered 1-3mg pills, each night, for up to 20 weeks
  Other Names: risperdal

SUMMARY:
The study aims to assess the efficacy and tolerability of risperidone added to lithium, valproate or lamotrigine in patients experiencing a manic episode with depressive or irritable features.

DETAILED DESCRIPTION:
* The study aims to assess the efficacy and tolerability of risperidone added to lithium, valproate or lamotrigine, or any combination of the three, in patients experiencing a manic episode with depressive or irritable symptoms.
* To assess the back ground and baseline features associated with response/non-response to risperidone plus mood stabilizer in patients with mania with depressive or irritable features.
* To assess the symptomatic dimensions of response of risperidone added to mood stabilizers in patients with mania with depressive or irritable features.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV diagnosis of bipolar disorder, currently manic, or mixed manic
* YMRS score>/= 16
* One or more of following:

  1. 3 MADRS depression items scoring >/=3
  2. 3 BISS depression items scoring >/=3
  3. YMRS irritability and aggressive items sum score>/=4
* Taking lithium, valproate or lamotrigine at stable dose for 4 wks or longer, with adequate serum level
* age 18 and over
* Male or female
* Inpatient or outpatient

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Forty percent reduction in YMRS | 20 weeks

SECONDARY OUTCOMES:
twenty percent reduction in MADRS | 20 weeks
Remission rate, defined as final score of plus or minus eight on YMRS and MADRS | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Singh, MD, Study Director — UT-SanAntonio; Charles Bowden, MD, Principal Investigator — UT San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States